CLINICAL TRIAL: NCT02203110
Title: The Impact of Simultaneous Presence of Viral and Bacterial Pathogens on Therapy and Course of Severe Pneumonia
Acronym: SCAHAVAP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: University of Ljubljana, Faculty of Medicine (Other)
Responsible Party: Principal Investigator, Primoz Karner, MD, University Medical Centre Ljubljana
Other Study IDs: Severe pneumonia
Record Dates: First submitted 2014-07-25; First posted 2014-07-29 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Community Acquired Pneumonia; Hospital Acquired Pneumonia; Ventilator Associated Pneumonia
Keywords: simultaneous bacterial and viral pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia; Healthcare-Associated Pneumonia; Pneumonia, Ventilator-Associated; Pneumonia, Viral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood, two 7 ml samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to determine if the clinical course of pneumonia is more severe when both, bacterial and viral pathogens are find as possible causative agent and how does it affect treatment.

DETAILED DESCRIPTION:
Basic demographic data of the patients (age, gender), data on concomitant diseases and epidemiological circumstances will be collected

Severity of illness will be assessed by APACHE II (at day 1) and SOFA (at day 1,2,3 and 7) scoring system

Following laboratory tests will be performed at day 1, 2,3 and 7.:

* blood count analysis
* differential blood count
* C- reactive protein, procalcitonin
* glucose, urea, potassium, sodium, chloride, magnesium, creatinine, bilirubin, protein, albumin, alkaline phosphatase, aspartate aminotransferase, alanine transaminase, gamma-glutamyl transpeptidase , alpha-amylase, lipase, creatine kinase, lactate dehydrogenase, myoglobin
* arterial blood gas analysis
* tests of hemostasis.

Additional 2 mL of blood will be taken at day 1 and day 21 (or later), due to paired serologic testing

To establish the presence of potential pathogens we will perform following microbiological investigations:

* cultivation of 2 pairs of blood cultures in all patients
* cultivation of sputum or quantitative cultivation of tracheal aspirate in nonintubated patients
* quantitative cultivation of tracheal aspirate or bronchoalveolar lavage in intubated patients
* testing the presence of soluble Legionella antigen in urine in all patients
* testing the presence of genetic material of respiratory viruses (influenza A, influenza B, respiratory syncytial virus , adenovirus, bocavirus, coronavirus, metapneumovirus, parainfluenza virus, rhinovirus) by qualitative polymerase chain reaction (PCR) in nasopharyngeal swabs in all patients, in the tracheal aspirate in nonintubated patients and in tracheal aspirate or bronchoalveolar lavage fluid in intubated patients
* testing the presence of mycoplasmal, legionella and chlamydial DNA by qualitative PCR in nasopharyngeal smears in all patients, in the tracheal aspirate in nonintubated patients and in bronchoalveolar lavage fluid or in tracheal aspirate in intubated patients

ELIGIBILITY:
Inclusion Criteria: diagnosis of

* severe community acquired pneumonia or
* severe hospital acquired pneumonia or
* ventilator--associated pneumonia

Exclusion Criteria:

* antibiotic treatment of actual episode of pneumonia for more than 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admited to Intensive Care Unit Department of Infectious Diseases University Medical Centre Ljubljana due to severe pneumonia or pneumonia will develop during their stay in ICU.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Rate of changes in empirical antibiotic therapy due to broad microbiological diagnostic | each patient will be assessed at enrollment and follow-up for 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Primoz Karner, Principal Investigator — Intensive Care Unit, Department of Infectious Diseases, University Medical Centre Ljubljana, Japljeva ulica 2, SI-1000 Ljubljana, Slovenia
Locations (1):
- Intensive Care Unit. Department of Infectious Diseases, Umiversity Medical Centre Ljubljana, Japljeva 2, Ljubljana, Slovenia